CLINICAL TRIAL: NCT02103569
Title: Effect of a Combination of Daclatasvir, Asunaprevir, and BMS-791325 on the Pharmacokinetics of a Combined Oral Contraceptive Containing Ethinyl Estradiol and Norethindrone Acetate in Healthy Female Subjects
Brief Title: Drug Interaction Study of an OCP (Norethindrone (ND) Acetate and Ethinyl Estradiol (EE))With a Combination of Daclatasvir (DCV) Asunaprevir (ASV) and BMS-791325
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: AI443-016
Record Dates: First submitted 2014-04-01; First posted 2014-04-04 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — asunaprevir; 8-cyclohexyl-N-((dimethylamino)sulfonyl)-1,1a,2,12b-tetrahydro-11-methoxy-1a-((3-methyl-3,8-diazabicyclo(3.2.1)oct-8-yl)carbonyl)cycloprop(d)indolo(2,1-a)(2)benzazepine-5-carboxamide; Ethinyl Estradiol; norethindrone acetate, ethinyl estradiol, ferrous fumarate drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1: FDC of NE/EE + DCV 3DAA FDC + BMS-791325 (Experimental): Cycle 1- Low dose FDC of Norethindrone and Ethinyl Estradiol tablet orally on specified days
  Cycle 2- High dose FDC of Norethindrone and Ethinyl Estradiol tablet orally on specified days and High dose FDC of Norethindrone and Ethinyl Estradiol + FDC of Daclatasvir, Asunaprevir and BMS-791325 + BMS-791325 tablets orally on specified days
  Interventions: Drug: FDC of Daclatasvir, Asunaprevir and BMS-791325; Drug: FDC of Norethindrone and Ethinyl Estradiol; Drug: BMS-791325

INTERVENTIONS:
Drug: FDC of Daclatasvir, Asunaprevir and BMS-791325
Drug: FDC of Norethindrone and Ethinyl Estradiol
  Other Names: Loestrin®
Drug: BMS-791325

SUMMARY:
The purpose of this study is to assess the effect of DCV/ASV/BMS-791325 fixed dose combination (FDC) + 75mg BMS-791325 on the Pharmacokinetics (PK) of the oral contraceptive agent.

DETAILED DESCRIPTION:
IND Number: 79,599 and 101,943

Other: Phase 1 Clinical Pharmacology drug interaction study in healthy female subjects

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Healthy females within age of 18-40 years
* Must be a Women of Childbearing potential
* Must be on a stable regimen of oral contraceptive therapy for at least 3 consecutive months prior to study start

Exclusion Criteria:

* Subjects must not have any significant acute or chronic medical illnesses or conditions precluding safe use of oral contraceptives
* Prior exposure to DCV, ASV or BMS-791325 within 30 days of dosing on study day 1
* Smoking within 6 months of study start

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Area under the concentration versus time curve in 1 dosing interval (AUC (TAU)) of Ethinyl Estradiol and Norethindrone | Day 21 to Day 49
Maximum observed plasma concentration (Cmax) of Ethinyl Estradiol and Norethindrone | Day 21 to Day 49

SECONDARY OUTCOMES:
Dose-normalized area under the concentration versus time curve in 1 dosing interval (AUC (TAU)) of Ethinyl Estradiol and Norethindrone | Day 1 to Day 50
Dose-normalized maximum observed plasma concentration (Cmax) of Ethinyl Estradiol and Norethindrone | Day 1 to Day 50
Time of maximum observed plasma concentration (Tmax) of Ethinyl Estradiol and Norethindrone | Day 1 to Day 50
Safety measured by occurrence of Adverse events (AEs), serious AEs and AEs leading to discontinuation | Day 1 to Day 50
Safety measured by abnormalities in vital sign measurements | Day 1 to Day 50
Safety measured by findings on Electrocardiogram (ECG) measurements and physical examinations | Day 1 to Day 50
Safety measured by marked abnormalities in clinical laboratory test results | Day 1 to Day 50

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Myers Squibb, Study Director — Bristol-Myers Squibb